CLINICAL TRIAL: NCT02391428
Title: The Correlation Between Blood omega3 and ADHD
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ayelet Omer Armon (Other Government)
Responsible Party: Sponsor-Investigator, Ayelet Omer Armon, Dr., Ziv Hospital
Organization: Ziv Hospital (Other Government)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ZIV-0019-14; Ziv (Other: medical center)
Record Dates: First submitted 2015-03-05; First posted 2015-03-18 (Estimated); Last update posted 2015-03-19 (Estimated); Status verified 2015-03

CONDITIONS: Attention Deficit Hyperactivity Disorder (ADHD)
Keywords: ADHD; omega3
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Hematologic Tests; Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Children who diagnosed with ADHD (Experimental): The ADHD children will be asked to consume omega3 capsules for 6 months. Blood will be taken for omega3 analysis in day 0, after 3 and 6 months.
  Interventions: Procedure: blood test; Dietary Supplement: omega3 capsules
- Control group of children without ADHD (Experimental): Blood test:
  The control group of 30 children (age and gender match) without ADHD and related neuropsychiatric syndromes, who were hospitalized due to surgical or orthopedic problems. Only when blood will be taken for clinical purposes, the investigators will ask the children and their parents to allow the collection of an additional small blood tube.
  Interventions: Procedure: blood test

INTERVENTIONS:
Procedure: blood test — Blood test: Small volume (3 ml) of blood will be taken by venipuncture into ethylenediaminetetraacetic acid (EDTA) tube.
Dietary Supplement: omega3 capsules — Only ADHD children will be given a supply of omega3 capsules (containing 400 mg EPA and 200 mg DHA)
  Arms: Children who diagnosed with ADHD

SUMMARY:
Attention deficit hyperactivity disorder (ADHD) is a major problem in children and adolescents. Clinical and biochemical evidence suggests that deficiencies of polyunsaturated fatty acids (PUFA) could be related to ADHD. PUFAs are the major components of brain with important physiologically active functions.

Aim: Study the relationship between omega3 blood values and ADHD clinical status.

Methods: The investigators will recruit 30 children, who have been diagnosed with ADHD by a child psychiatrist. In addition the investigators will recruit a control group of 30 children without ADHD and related neuropsychiatric syndromes. Blood will be taken from all children.

The ADHD children will be asked to consume omega3 capsules for 6 month. After 3 and 6 months, all children will undergo clinical examination and blood tests will be taken for omega3 index analysis. Blind frozen samples of isolated red blood cell (RBC) will be analyzed according to the omega3 index methodology.

DETAILED DESCRIPTION:
Attention deficit hyperactivity disorder (ADHD) is a major problem in children and adolescents. Clinical and biochemical evidence suggests that deficiencies of polyunsaturated fatty acids (PUFA) could be related to ADHD. PUFAs are the major components of brain with important physiologically active functions.

Aim: To investigate influence effects of omega3 dietary supplementation on ADHD symptoms and the measured blood values.

Methods: The study will be authorized by the Ziv Helsinki Committee and the Ministry of Health. Written Informed consent will obtained from parents. The investigators will recruit 30 children, who have been diagnosed with ADHD by a child psychiatrist. In addition the investigators will recruit a control group of 30 children without ADHD and related neuropsychiatric syndromes. Blood will be taken from all children.

ELIGIBILITY:
Inclusion Criteria:

- ADHD group: Children diagnosed with ADHD aged 6-14; children who have not received a dietary supplement of omega3 in the last month

Control group inclusion criteria: Children without ADHD and related neuropsychiatric syndromes aged 6-14, Children who have not received a dietary supplement of omega3 in the last month.

Exclusion Criteria:

- Children with severe chronic or autoimmune disorders, children who received a dietary supplement of omega3 in the last month

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2015-04; Primary Completion 2015-09 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
blood omega3 | 6 month

SECONDARY OUTCOMES:
ADHD Symptoms | 6 month
  Will be assessed using the ADHD Rating Scale IV (ADHD RS).